CLINICAL TRIAL: NCT00734136
Title: Role Of Angiogenic Factors In The Development Of Hepatorenal Syndrome
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient findings for data analysis
Sponsor: Lahey Clinic (Other)
Collaborators: Beth Israel Deaconess Medical Center (Other); Dr. Vikas Sukhatme (Unknown)
Responsible Party: Mary Ann Simpson, Ph.D., Lahey Clinic, Inc.
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2005-040
Record Dates: First submitted 2008-08-12; First posted 2008-08-14 (Estimated); Last update posted 2009-02-18 (Estimated); Status verified 2009-02

CONDITIONS: Hepatorenal Syndrome; Renal Failure; Liver Diseases
Keywords: Angiogenic Factors; Hepatorenal Syndrome; Liver Disease; Renal Failure; Liver Cirrhosis; Ascites
MeSH Terms: conditions — Hepatorenal Syndrome; Renal Insufficiency; Liver Diseases; Liver Cirrhosis; Ascites | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Other): 50 surgical subjects undergoing either liver transplantation or hepatic resection
  Interventions: Procedure: Blood Draws and a hepatectomy specimen
- 2 (Other): 50 Subjects with Liver disease who are are not surgical candidates
  Interventions: Procedure: Blood draw - pre operative standard of care

INTERVENTIONS:
Procedure: Blood Draws and a hepatectomy specimen — Pre operative blood draw(1.5 ml serum, 1.5 ml EDTA)(approximately 2 teaspoons).
  Blood draw during surgery(1.5 ml serum, 1.5 ml EDTA)from Hepatic Artery, Hepatic Vein, and Portal Vein.
  Wedge section of Hepatectomy specimen following resection in surgical subjects(tested for the same factors)
  Arms: 1
Procedure: Blood draw - pre operative standard of care — Pre-operative blood draw(1.5 ml serum, 1.5 ml EDTA)(approximately 2 teaspoons) from peripheral vein
  Arms: 2

SUMMARY:
This Study will look at the effect of substances called "angiogenic factors"(development of new blood vessels) have on the development of severe liver disease. The results may help to understand the factors involved in the repair and regeneration of liver tissue and to see if different types of liver disease are associated with different types of factors, especially in the severe liver disease called hepatorenal syndrome.

DETAILED DESCRIPTION:
Renal dysfunction in patients who also suffer from end stage liver disease is associated with increased morbidity and mortality comparted to patients suffering from liver disease alone. If frank renal failure develops in a patient with cirrhosis and ascites, the median survival time from onset of renal failure is approximately 2 weeks. Kidney dysfunction may be transient, secondary to pooling of blood in the splanchnic bed and consequent reduction in renal blood flow. In this instance, liver transplantation and restoration of normal circulatory patterns will result in return of normal renal function.

Currently, there is no diagnostic test to differentiate between temporary and permanent renal dysfunction in the presence of end stage liver disease. As a result, the number of combined liver-kidney transplant occuring has steadily increased. Slightly more than 20%(8 of 38) of the liver transplants performed by our service in 2004 have been combined liver-kidney transplants. The double procedure increases the length of anesthesia exposure and surgical time, and the presence of the transplanted kidney may require increased immunosuppression in comparison to a liver-only transplant.

We plan to examine the role of angiogenic factors in the abnormal blood flow patterns known to be associated with hepatorenal syndrome.

Specimen analysis: Circulating levels of cytokines and growth factors will be measured using commercially available ELISAs. Matrix metalloproteins will be measured by quantitative electrophoresis.

Expression of A20 will be determined by extraction of total RNA from whole blood using Trizol and run in standard Northern blot methodology. RNA will by hybridized with [³²P]-dATP labeled A20 probes and glyceraldehyde-3-phosphate dehydrogenase(GAPDH) or β-actin probes to correct for uneven loading. Similar RNA extraction will be performed on liver tissue obtained at time of surgery. Microarray analysis will be performed on the extract to identify specific genes that may be involved in the pathogenesis of HRS.

Results of laboratory analyses will be correlated with clinical parameters and attempts will be made to identify specific cytokines or up-regulated genes with particular phases or degree or renal dysfunction in patients with liver disease. Similar analyses will be performed in patients with other types of hepatic disease.

ELIGIBILITY:
Inclusion Criteria:

* Sign informed consent
* Subjects who present for Liver Transplantation
* Subjects who present for Hepatic resection
* Subjects with Non-Surgical Liver Disease

Exclusion Criteria:

* Absence of Liver Disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2005-05; Primary Completion 2005-07 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Analysis of Blood samples for angiogenic factors | 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Mary Ann Simpson, Ph.D., Principal Investigator — Lahey Clinic, Inc.
Locations (1):
- Lahey Clinic, Inc., Burlington, Massachusetts, United States

REFERENCES:
- [Background] Levine RJ, Maynard SE, Qian C, Lim KH, England LJ, Yu KF, Schisterman EF, Thadhani R, Sachs BP, Epstein FH, Sibai BM, Sukhatme VP, Karumanchi SA. Circulating angiogenic factors and the risk of preeclampsia. N Engl J Med. 2004 Feb 12;350(7):672-83. doi: 10.1056/NEJMoa031884. Epub 2004 Feb 5. PMID 14764923